CLINICAL TRIAL: NCT01681667
Title: Tablet vs. Liquid Suspension Ibuprofen in the Relief of Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Wayne Triner, Professor and Research Director Dept.of Emergency Medicine, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3003
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Pharyngitis
MeSH Terms: conditions — Pharyngitis | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ibuprofen (Active Comparator): liquid ibuprofen 400mg compared to tablet ibuprofen 400mg
  Interventions: Drug: Ibuprofen
- sugar pill or liquid (Placebo Comparator)

INTERVENTIONS:
Drug: Ibuprofen — ibuprofen liquid 400mg vs. ibuprofen tablet 400mg
  Arms: ibuprofen

SUMMARY:
Ibuprofen (also known as Advil or Motrin) is a medication that is known to reduce pain. It is also known that ibuprofen levels in the blood rise higher and faster if the medication is taken in liquid suspension. This study will attempt to determine if ibuprofen suspended in a liquid works to relieve sore throat pain faster than pills of ibuprofen. It will also determine whether patients with sore throat prefer to take pill or liquid form of the medication.

DETAILED DESCRIPTION:
Pain is a common emergency and urgent care complaint. Ibuprofen is known to be an effective treatment for many forms of pain. Sore throat has been established to be an acceptable model of analgesic effect, and ibuprofen has been found to offer relief in studies of sore throat. Several studies have demonstrated that ibuprofen in suspension is absorbed into the system more quickly and results in earlier maximum blood concentrations. To date, no study has evaluated onset to analgesia as reported by the patient for suspension versus tablet formation of ibuprofen in an emergency department population presenting with complaints of sore throat. This is a double blinded randomized placebo controlled trial to compare suspension versus tablet ibuprofen in an emergency department population presenting with sore throat. The purpose of this study is to assess whether ibuprofen in suspension form results in relief of pain more quickly than the tablet form of an equivalent dose of ibuprofen. We will also determine if there is an interval difference from time of analgesia administration to perception of analgesia that is clinically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 12 years and less than 65 years
* Weight > 40 kg
* a provider order for ibuprofen to address pharyngitis pain.
* Initial Numeric Pain Score > 6

Exclusion Criteria:

* Known allergy or hypersensitivity to aspirin or NSAIDs
* Inability to swallow pills
* Inability to carry out informed consent in English
* Inability to complete a visual analog pain scale
* A concomitant order for another class of analgesic
* Use of analgesic within 8 hours
* Known 3rd trimester pregnancy
* Significant medical conditions where participation would pose an unnecessary barrier to ongoing care.
* Those taking opioid medications for more than 3 days
* Weight < 40 kg

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Time of pain relief | 1 hour
  Comparing liquid ibuprofen to tablet ibuprofen to determine which works faster to relieve sore throat pain. We will also determine whether patients with sore throat prefer to take pill or liquid form of medication.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne R Triner, DO, MPH, Principal Investigator — Albany Medical College Department of Emergency Medicine
Locations (1):
- Albany Medical Center Emergency Department, Albany, New York, United States